CLINICAL TRIAL: NCT05817188
Title: Translational Identification of Medication Repurposing Candidates to Slow Cognitive Decline in Dementia
Brief Title: Medication Repurposing to Stop Cognitive Decline in Dementia
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: KTH Royal Institute of Technology (Other); Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Sara Garcia-Ptacek, Assistant Professor/Docent (title formerly translated Assoc Prof), Karolinska Institutet
Other Study IDs: 2022-01425
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2023-04

CONDITIONS: Alzheimer Dementia; Dementia Disorders
Keywords: medication; repurposing; cognitive decline; dementia; Mini-Mental State Examination
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Dementia patients: This register-based project will include all patients diagnosed with dementia and registered in the Swedish Registry for Cognitive/Dementia Diseases. Identification of cases and control and data collation are carried out by Swedish authorities.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention was applied

SUMMARY:
Dementia creates a great personal and societal burden and there are currently no treatments to stop memory loss. Many patients with dementia take medications to treat other conditions, e.g. high blood pressure and cholesterol. Some of these medications may have central effects on the pathophysiological processes leading to dementia.

Medication repurposing is a cost and time-effective way to discover new treatments. Swedish registers are a unique tool to detect medication candidates for repurposing. The Swedish Dementia Registry (SveDem) has >100000 patients and ca. 144000 measures of cognition over time (measured with the Mini-Mental State Examination-MMSE), making it perfect to examine whether certain medications are associated with less cognitive decline in patients with dementia. Cholesterol and kidney function affect treatment and cognition and are available for 25000 patients. The investigators propose a study combining traditional cohort studies and newer artificial intelligence (machine learning) techniques to detect medications associated with slower cognitive decline in patients from SveDem. The investigators will test pre-specified hypotheses since the investigators suspect specific medications are better candidates to prevent cognitive decline, but the investigators will also let the machine learning algorithms explore the data to find associations that the investigators do not suspect in advance. Finally, the candidate medications will be tested in animal and cellular models to determine the mechanisms of their effects.

ELIGIBILITY:
Inclusion Criteria:

All patients with dementia registered in SveDem.

Exclusion Criteria:

Lack of Swedish personal identification number or coordination number.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes >100,000 patients in SveDem and ca. 144,000 measures of Mini-mental State Examination (MMSE) including base registration and follow-ups. Our current merged dataset contains 80,004 individuals, but we periodically conduct new merges which will increase the sample size in the future: this may be necessary for rarer medications.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Cognitive decline | Through study completion, at least 1 year
  The data on cognitive decline will be assessed by Mini Mental State Examination (MMSE) score. The MMSE score ranges from 0 and 30. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Rate of nursing home placement | Through study completion, at least 1 year
  Data will be obtained from the social services registry.
Mortality | Through study completion, at least 1 year
  Data about date and cause(s) of death will be collected from The Cause of Death Register.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Garcia-Ptacek, MD,PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Religa D, Fereshtehnejad SM, Cermakova P, Edlund AK, Garcia-Ptacek S, Granqvist N, Hallback A, Kawe K, Farahmand B, Kilander L, Mattsson UB, Nagga K, Nordstrom P, Wijk H, Wimo A, Winblad B, Eriksdotter M. SveDem, the Swedish Dementia Registry - a tool for improving the quality of diagnostics, treatment and care of dementia patients in clinical practice. PLoS One. 2015 Feb 19;10(2):e0116538. doi: 10.1371/journal.pone.0116538. eCollection 2015. PMID 25695768
- [Background] Garcia-Ptacek S, Kareholt I, Farahmand B, Cuadrado ML, Religa D, Eriksdotter M. Body-mass index and mortality in incident dementia: a cohort study on 11,398 patients from SveDem, the Swedish Dementia Registry. J Am Med Dir Assoc. 2014 Jun;15(6):447.e1-7. doi: 10.1016/j.jamda.2014.03.001. Epub 2014 Apr 8. PMID 24721339
- [Background] Roheger M, Zupanic E, Kareholt I, Religa D, Kalbe E, Eriksdotter M, Garcia-Ptacek S. Mortality and nursing home placement of dementia patients in rural and urban areas: a cohort study from the Swedish Dementia Registry. Scand J Caring Sci. 2018 Dec;32(4):1308-1313. doi: 10.1111/scs.12574. Epub 2018 Apr 14. PMID 29656469
- [Background] Garcia-Ptacek S, Modeer IN, Kareholt I, Fereshtehnejad SM, Farahmand B, Religa D, Eriksdotter M. Differences in diagnostic process, treatment and social Support for Alzheimer's dementia between primary and specialist care: resultss from the Swedish Dementia Registry. Age Ageing. 2017 Mar 1;46(2):314-319. doi: 10.1093/ageing/afw189. PMID 27810851
- [Background] Cermakova P, Nelson M, Secnik J, Garcia-Ptacek S, Johnell K, Fastbom J, Kilander L, Winblad B, Eriksdotter M, Religa D. Living Alone with Alzheimer's Disease: Data from SveDem, the Swedish Dementia Registry. J Alzheimers Dis. 2017;58(4):1265-1272. doi: 10.3233/JAD-170102. PMID 28550260
- [Background] Garcia-Ptacek S, Kareholt I, Cermakova P, Rizzuto D, Religa D, Eriksdotter M. Causes of Death According to Death Certificates in Individuals with Dementia: A Cohort from the Swedish Dementia Registry. J Am Geriatr Soc. 2016 Nov;64(11):e137-e142. doi: 10.1111/jgs.14421. Epub 2016 Nov 1. PMID 27801938
- [Background] Mo M, Abzhandadze T, Hoang MT, Sacuiu S, Jurado PG, Pereira JB, Naia L, Kele J, Maioli S, Xu H, Eriksdotter M, Garcia-Ptacek S. Antidepressant use and cognitive decline in patients with dementia: a national cohort study. BMC Med. 2025 Feb 25;23(1):82. doi: 10.1186/s12916-025-03851-3. PMID 39994788
- [Background] Grau-Jurado P, Mostafaei S, Xu H, Mo M, Petek B, Kalar I, Naia L, Kele J, Maioli S, Pereira JB, Eriksdotter M, Chatterjee S, Garcia-Ptacek S. Medications and cognitive decline in Alzheimer's disease: Cohort cluster analysis of 15,428 patients. J Alzheimers Dis. 2025 Feb;103(3):931-940. doi: 10.1177/13872877241307870. Epub 2025 Jan 8. PMID 39772858
- [Background] Petek B, Habel H, Xu H, Villa-Lopez M, Kalar I, Hoang MT, Maioli S, Pereira JB, Mostafaei S, Winblad B, Gregoric Kramberger M, Eriksdotter M, Garcia-Ptacek S. Statins and cognitive decline in patients with Alzheimer's and mixed dementia: a longitudinal registry-based cohort study. Alzheimers Res Ther. 2023 Dec 20;15(1):220. doi: 10.1186/s13195-023-01360-0. PMID 38115091
- See also: Related Info — http://www.svedem.se